CLINICAL TRIAL: NCT06450704
Title: Inflammatory and Brain Mechanisms and Clinical and Cognitive Effects of an Exercise Intervention in Major Depressive Disorder: a Randomised Longitudinal Clinical Trial.
Brief Title: Cerebral and Anti-inflammatory Response Through Exercise - Mechanisms In Depressive Disorders
Acronym: CARE-MIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Principe de Asturias (Other); Quirón Madrid University Hospital (Other); Universidad Autonoma de Madrid (Other); Centro de Investigación Biomédica en Red de Salud Mental (Network); Hospital Universitario Puerta de Hierro de Majadahonda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5561
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Inflammatory Response
Keywords: Major Depressive Disorder; Physical Exercise; Inflammation; Neuroimaging
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity; Inflammation | interventions — Exercise; Exercise Therapy; Antidepressive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (EG) (Experimental): Major Depressive Disorder patients will receive the exercise intervention for 12 weeks as an add-on to their usual treatment (antidepressant treatment prescribed by the attending specialist). They will gradually increase their levels of physical activity by daily walking and will conduct aerobic and muscle strength activities 2 days per week. The program will be supervised by a physical education and sports professional.
  Interventions: Other: Physical Exercise; Drug: Antidepressant medication (ADM)
- Control group (CG) (Active Comparator): Major Depressive Disorder patients will only receive standard treatment (antidepressant treatment prescribed by the attending specialist) and will be instructed to not change their usual physical activity.
  Interventions: Drug: Antidepressant medication (ADM)

INTERVENTIONS:
Other: Physical Exercise — Daily walking. Participants will be given an activity band to self-monitor the number of steps they walk each day during the 12-week intervention period. Each participant must reach a certain number of daily steps with a progressive goal adjusted to the number of steps from the previous week. The goal is set considering the superior number to the median of steps of the preceding week.
  Weekly combined exercise sessions (aerobic + strength exercise) 2 sessions of 60 minutes per week in a 12-week program. The exercise intervention will combine the use of elastic bands and the body weight. First, 5 minutes of warm-up; second, training circuit with low-intensity strength exercises alternating work and rest times using rhythmic music. Upper, lower and middle body exercises will alternate. The program will progress in intensity, work: rest ratio, and technical difficulty of the exercises. At the end of the main part, there will be a cool-down and stretching for 5 minutes.
  Other Names: Therapeutic Exercise; physical activity; Exercise
  Arms: Exercise intervention group (EG)
Drug: Antidepressant medication (ADM) — Patients will receive their standard antidepressant treatment prescribed by their psychiatrist.

SUMMARY:
The goal of this clinical trial is to study how physical exercise works when applied to patients diagnosed with Major Depressive Disorder (MDD). The main questions it aims to answer are:

* What are the antiinflammatory and oxidative stress and neural mechanisms involved in the antidepressant effects of exercise?
* How effective is a physical exercise program in MDD patients in real-life conditions?

The experimental group will receive an exercise intervention as an add-on to their usual treatment (antidepressant treatment prescribed by the attending specialist). Researchers will compare to a control group, which will only receive standard treatment (antidepressant treatment prescribed by the attending specialist) and will be instructed to not change their usual physical activity. The aim is to see if a physical exercise intervention would induce a significant improvement in depressive symptoms and which mechanisms are responsible for this result.

DETAILED DESCRIPTION:
RATIONALE, BACKGROUND AND CURRENT STATUS

Although it is well established that physical exercise (PE) is efficacious in treating mild to moderate depression [1], it remains underprescribed and there are large gaps in knowledge of the neurobiological mechanisms involved in the antidepressant effect of physical exercise. Depression is a common and disabling illness, affecting over 300 million people worldwide. Despite existing effective treatments for MDD, half of patients exhibit recurrences and about one-third are resistant to treatment [2]. Therefore there is an important need for new conceptual frameworks for understanding the pathophysiology of depression and for the implementation of cost-effective, acceptable to patients and feasible augmentation strategies for the treatment of MDD.

The underlying neurobiological mechanisms for exercise-related clinical improvement in depression remain understudied and require further investigation. From a physiological perspective, converging evidence suggests that exercise and antidepressant medication may alleviate depression through common neuromolecular mechanisms, including reduced inflammatory signalling [3] and increased expression of neuroplasticity [4]. There is substantial evidence about the contribution of low-grade inflammatory mechanisms to the pathophysiology of depression [5-7]. Increases in inflammation can elicit depression symptoms such as sad mood, anhedonia, fatigue, psychomotor retardation, and social-behavioural withdrawal [8].

Increasing evidence indicates that exercise exerts many benefits through activating Nrf2 signalling [9]. Nrf2 is a key master transcription factor that controls the expression of over 100 anti-oxidative and anti-inflammatory genes and that is dysfunctional in preclinical studies of depression. [10]. The protective effects of exercise are not seen when Nrf2 is blocked, supporting the role of Nrf2 in exercise-mediated neuroprotection [9]. To date, no exercise intervention studies have been conducted on Nrf2 signaling in humans.

There is a significant gap in the literature regarding the anti-inflammatory properties of exercise as add-on to antidepressant treatment. Well-conducted and more extensive studies are necessary to confirm any additive or synergistic effects between antidepressant drugs and physical exercise on inflammatory markers in MDD patients and its clinical relevance to treatment success or recurrence of MDD.

HYPOTHESIS

1. A physical exercise intervention as add-on to the conventional treatment of MDD will lead to antiinflammatory effects and less oxidative stress via Nrf2.
2. The exercise intervention would induce functional and structural changes in the brain of MDD patients treated with combined exercise and standard treatment.

3.12 weeks of an exercise intervention in real-life conditions would lead to a significant better outcome of depressive symptoms (Hamilton depression rating scale) in MDD patients treated with combined exercise and standard treatment compared to MDD patients treated only with standard treatment.

4. A 12-week exercise intervention will be associated with significantly greater improvements in cognitive performance than standard treatment alone.

5. A 12-week exercise intervention will be associated with significantly greater improvements in functioning and well-being than standard treatment alone.

6. One year after the exercise intervention, there will remain antidepressant and procognitive effects.

7. The combination of physical exercise to the standard treatment of MDD will be better accepted by patients than standard treatment alone.

8. Increase in awareness and skills of health practitioners on the antidepressant effect of exercise will lead to the incorporation of exercise prescription into clinical practice.

AIMS

This project aims to:

1. Analyze the effects of physical exercise on inflammation and oxidative stress, studying the activity levels of Nrf2 before and after the exercise intervention in MDD patients.
2. Study volumetric changes and cortical thickness, structural and functional connectivity and microstructural changes in the white matter in the brain after a 12-week exercise intervention.
3. Compare the antidepressant effect of a 12-week exercise intervention in real-life conditions combined with standard treatment to standard treatment and to study the change in symptom severity after the exercise intervention.
4. Explore changes in the cognitive performance of MDD patients after a 12-week exercise intervention.
5. Assess functioning and well-being after a 12-week exercise intervention in MDD patients.
6. Investigate if the clinical and cognitive changes persist 1 year after the beginning of the exercise intervention.
7. Evaluate the patient´s acceptability of an exercise-based intervention.
8. Increase awareness and skills of health practitioners on the anti-depressive effect of exercise.

DESIGN

It is proposed to carry out a multicenter, randomised, two-arm, parallel assignment, prospective, controlled trial of 12 weeks of exercise intervention, that includes a follow-up period of 1 year post-randomization.

Study arms:

1. Exercise intervention group (EG): MDD patients will receive the exercise intervention as an add-on to their usual treatment (antidepressant treatment prescribed by the attending specialist).
2. Control group (CG): MDD patients will only receive standard treatment (antidepressant treatment prescribed by the attending specialist) and will be instructed to not change their usual physical activity.

Eligible patients will be randomly allocated (1:1) to the study arms, using a block randomization scheme. The exercise intervention will last 12 weeks and subjects will be assessed at 3-time points: at baseline before the randomization (T0); 12 weeks after the beginning of the intervention (T1) and 1 year after randomization (T2). The evaluation of the effect of the intervention will be blind. The clinical researchers that will assess patients at T1 and T2 will not know if the patients have been assigned to the EG or the CG. Patients will be instructed not to disclose their participation in the exercise program to the evaluators.

Exercise intervention

The exercise intervention program in real-life conditions will consist of two components:

1. to gradually increase the levels of physical activity by daily walking
2. additionally, participants will conduct aerobic and muscle strength activities 2 days per week. The program will be supervised by a physical education and sports professional with more than 10 years of experience in promoting physical exercise in MDD and several mental disorders patients.

Daily walking: Participants will be given an activity band (MiBand6) to self-monitor the number of steps they walk each day during the 12-week intervention period. The number of steps will be recorded with the activity band Miband6 and will automatically be sent to the exercise coach through the proper activity band configuration. The goal is set considering the superior number to the median of steps of the preceding week.

Weekly combined exercise sessions (aerobic + strength exercise): Participants will be scheduled to participate in 60-minute supervised online group sessions twice per week in a 12-week program. The exercise intervention will combine the use of elastic bands and the body weight. The exercise coach will supervise the exercise through a virtual connection allowing technical corrections and checking the proper performance of the activity. After 5 minutes of warm-up, the main part will begin, which consists of a training circuit with low-intensity strength exercises alternating work and rest times using rhythmic and melodic music preferred by the participants. Upper, lower and middle body exercises will alternate. The program will progress in intensity (using more resistant bands), work: rest ratio (starting at 30:30 and ending at 45:15), and technical difficulty of the exercises. At the end of the main part, there will be a cool-down and stretching for 5 minutes.

The effectiveness of this physical activity intervention will be assessed through:

1. Online supervision twice a week by a physical education and sports professional during the combined exercise sessions. Additionally, this professional will receive the number of steps the participants have walked every day of the week through the activity band Miband6 and will send a weekly message to the participants to propose an individualized goal of steps for the upcoming week.
2. Movement-related behaviours (i.e., physical activity, sedentary behaviour, and sleep time) will be measured by the wrist-worn tri-axial accelerometer ActiGraph GT9X Link (Pensacola, FL, USA). The accelerometer will be worn 24 hours over 7 days at the onset of the exercise intervention and 7 days post-intervention. Sleep time, sedentary activity, and mild and moderate-intense physical activity will be objectively estimated using the data monitored by multiple sensors and using specific algorithms (ActiLife software v6.13.4; ActiGraph Corp., LLC).

STUDY SUBJECTS

A total of 124 MDD patients will be enrolled across a 3 year period. Patients' recruitment will be done in 4 participating centres in the region of Madrid (N=31 in each participating centre): Hospital La Princesa, Hospital La Paz, Hospital Ramón y Cajal and Hospital Principe de Asturias. All centres will follow the same research protocol.

ANALYSES

Differences between and within groups for continuous variables in the change from baseline to endpoint (12 weeks) and data concerning the 3-time points (baseline, 12 weeks, 1 year) will be analysed using a repeated-measurement, likelihood-based mixed-effect model with an unstructured variance matrix. Dichotomous variables will be assessed with odds ratios and χ2 tests. Potential moderators of the intervention will be examined by testing interaction terms between the intervention group and baseline characteristics (age, gender, clinical centre, treatment and baseline levels of BMI and physical activity). A generalised linear mixed model will be used to study changes over time in the study variables (clinical, cognitive, and biological biomarkers). Multiple regression models will be performed to explore predictive variables associated with clinical or cognitive changes. Confounding variables (concomitant pharmacological treatment and regular physical activity) will be controlled in the regression model. A compositional data analysis will be performed to explore associations between variables of interest and the composition of activity using multiple lineal regression models. All analyses will follow the intent-to-treat (ITT) principle. Statistical analyses will be performed using the IBM SPSS statistical software package (v.24.0, Chicago, IL, USA) and R software. The significance level will be set at P<0.05 and the confidence intervals will be calculated at 95%.

SAMPLE SIZE AND POWER ANALYSIS

Based on previous studies [11], a two-sided type 1 error probability of 5% with a Bonferroni adjusted α of .05/2 = .025 to allow for comparison of the 2 arms of the trial, as well as a minimal clinically relevant difference of 5 points on the Ham-D17, a standard deviation of 5.5 points, a β= .20 (power of 80%), and an anticipated dropout rate of 17% [12], we calculated that we needed a minimum of 124 patients (n=62/study arm), to detect clinically meaningful antidepressive changes after the physical exercise intervention.

LIMITATIONS

The study is designed as an add-on to usual MDD treatment which allows the apply a real-life conditions approach and will favour the transference of the results, however, the independent effect of exercise will not be assessed. For the same reason and to increase recruitment, homogeneity in the baseline pharmacological treatment will not be possible. An ideal design would select patients with similar severity characteristics to ascertain the clinical effect of exercise. However, it would limit the sample size and lead to an underpowered trial. This ecological approach would allow transference to clinical practice and acceptability by patients.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Major Depressive Disorder (MDD) according to DSM-5 criteria (through the Mini International Neuropsychiatric Interview (MINI)
* Severity of depression according to the Hamilton Depression Rating Scale 17 items (HAM-D17): minimum of 14 cut-off score of moderate depression.
* Outpatient clinical care.
* Current antidepressant treatment that will be maintained during the 12 weeks of the physical exercise intervention.

Exclusion Criteria:

* Diagnosis of any axis I diagnosis except for MDD;
* Contraindications for Magnetic Resonance Imaging.
* Antiinflammatory treatments or antibiotics within the week before randomisation.
* Vaccines within the month before randomisation.
* Fever (>38ºC) at the moment of study entry.
* Pregnant women.
* Alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory and oxidative stress biomarkers | 1. Before randomization; 2. 12-weeks after the beggining of intervention; 3. 1 year after randomization
  Nrf2 activity will be measured in circulating monocytes and through transcriptomic analysis of redox and inflammation related genes. Plasma levels of hs C-reactive protein (CRP), interleukin 6 (hs-IL-6) and tumoral nechrosis factor alfa (hs- TNF-alfa) will be analyzed.
Brain imaging | 1. Before randomization; 2. 12 Weeks after the beggining of intervention
  It will be evaluated using Magnetic Resonance Imaging. Four different sequences will be acquired: a) a T2-FLAIR sequence; b) a 3D T1w MPRAGE sequence; c) a Diffusion Weighted sequence and d) a T2 resting-state sequence. These data will be used to discard any neurological issues, to evaluate structural changes, and for other images coregistration, to evaluate the integrity of white matter and structural connectivity, and to evaluate functional connectivity.
Clinical evaluation | 1. Before Randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  The change in depression symptoms will be measured with the HAM-D17 scale. Duration of illness, number of episodes, current treatments, resistance antidepressant treatment index (Thase) will also be assessed.

SECONDARY OUTCOMES:
Cognitive evaluation | 1. Before Randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  Learning and verbal memory through the Hopkins Verbal Learning Test-Revised (HVLT-R); executive functioning through the Trail Making Test part B (TMT-B); processing speed through the Salthouse Perceptual Comparison Test (SPCT).
Functioning and Well-Being | 1. Before randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  The patient's functioning will be assessed through the WHO-DAS-II and well-being will be measured with the Cantrill ladder.
Muscle strength | 1. Before randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  It will be directly measured through a handheld dynamometer (TKK 5401 Grip-D, Takey, Tokyo, Japan) and a dynamometer for the upper and lower extremities (Lafayette Instruments dynamometer, Lafayette, Ind).
Cardiorespiratory fitness | 1. Before randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  It will be measured using the Incremental Shuttle Walk Test with blood gas analysis. The Incremental Shuttle Walk Test is performed on a flat 10-meter course marked by two cones. Participants are guided by auditory stimuli, which indicate when to increase speed (three beeps) and change direction at the end of the course (one beep). The test ends when the participant is more than 0.5 meters from the cone when the beep sounds (twice consecutively), reports being too short to continue, or experiences some discomfort that prevents them from continuing.
24-hours physical activity behaviors | 1. Before Randomization; 2. 12 Weeks after the beggining of intervention
  Physical activity, sedentary behaviour, and sleep will be objectively measured using a multi-sensor monitor (ActiGraph GT9X Link, Pensacola, FL, USA) over a 24-hour period, both at the onset of the exercise intervention and 7 days post-intervention. Only participants who carry the monitor for at least 95% of the day (1368 minutes) will be included in the analysis. This monitor is worn as a watch and will be placed on the non-dominant wrist.
  The Simple Physical Activity Questionnaire (SIMPAQ) will also be used as a self-reported measure of physical activity.
  Daily steps will be recorded through the activity band (MiBand6).
Anthropometric evaluation | 1. Before randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  Weight will be assessed through a stadiometer (SECA) and waist circumference with a metric tape (Harpenden anthropometric tape, Holtain Ltd). Body Mass Index, waist-to-hip ratio and blood pressure also will be assessed.
Metabolic biomarkers | 1. Before randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  Serum levels of glucose, glycosylated haemoglobin and lipid profile.
Nutrition habits | 1. Before randomization; 2. 12 Weeks after the beggining of intervention; 3. 1 Year after randomization
  It will be assessed with the Food Frequency Questionnaire (FFQ).

CONTACTS AND LOCATIONS:
Overall Officials: Pilar López García, PhD, Principal Investigator — Universidad Autonoma de Madrid
Locations (5):
- Spain (5):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravindran AV, Balneaves LG, Faulkner G, Ortiz A, McIntosh D, Morehouse RL, Ravindran L, Yatham LN, Kennedy SH, Lam RW, MacQueen GM, Milev RV, Parikh SV; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 5. Complementary and Alternative Medicine Treatments. Can J Psychiatry. 2016 Sep;61(9):576-87. doi: 10.1177/0706743716660290. Epub 2016 Aug 2. PMID 27486153
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Mathur N, Pedersen BK. Exercise as a mean to control low-grade systemic inflammation. Mediators Inflamm. 2008;2008:109502. doi: 10.1155/2008/109502. Epub 2009 Jan 11. PMID 19148295
- [Background] Dishman RK, Berthoud HR, Booth FW, Cotman CW, Edgerton VR, Fleshner MR, Gandevia SC, Gomez-Pinilla F, Greenwood BN, Hillman CH, Kramer AF, Levin BE, Moran TH, Russo-Neustadt AA, Salamone JD, Van Hoomissen JD, Wade CE, York DA, Zigmond MJ. Neurobiology of exercise. Obesity (Silver Spring). 2006 Mar;14(3):345-56. doi: 10.1038/oby.2006.46. PMID 16648603
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486
- [Background] Miller AH, Raison CL. The role of inflammation in depression: from evolutionary imperative to modern treatment target. Nat Rev Immunol. 2016 Jan;16(1):22-34. doi: 10.1038/nri.2015.5. PMID 26711676
- [Background] Slavich GM, Irwin MR. From stress to inflammation and major depressive disorder: a social signal transduction theory of depression. Psychol Bull. 2014 May;140(3):774-815. doi: 10.1037/a0035302. Epub 2014 Jan 13. PMID 24417575
- [Background] Zuo C, Cao H, Song Y, Gu Z, Huang Y, Yang Y, Miao J, Zhu L, Chen J, Jiang Y, Wang F. Nrf2: An all-rounder in depression. Redox Biol. 2022 Dec;58:102522. doi: 10.1016/j.redox.2022.102522. Epub 2022 Oct 31. PMID 36335763
- [Background] Done AJ, Traustadottir T. Nrf2 mediates redox adaptations to exercise. Redox Biol. 2016 Dec;10:191-199. doi: 10.1016/j.redox.2016.10.003. Epub 2016 Oct 14. PMID 27770706
- [Background] Krogh J, Saltin B, Gluud C, Nordentoft M. The DEMO trial: a randomized, parallel-group, observer-blinded clinical trial of strength versus aerobic versus relaxation training for patients with mild to moderate depression. J Clin Psychiatry. 2009 Jun;70(6):790-800. doi: 10.4088/jcp.08m04241. PMID 19573478
- [Background] Stubbs B, Vancampfort D, Rosenbaum S, Ward PB, Richards J, Soundy A, Veronese N, Solmi M, Schuch FB. Dropout from exercise randomized controlled trials among people with depression: A meta-analysis and meta regression. J Affect Disord. 2016 Jan 15;190:457-466. doi: 10.1016/j.jad.2015.10.019. Epub 2015 Oct 29. PMID 26551405